CLINICAL TRIAL: NCT02289924
Title: PERSEUS-IT. A Prospective Non-intERventional Study to asSEss the Effectiveness of Aflibercept (Eylea®) in roUtine Clinical Practice in patientS With Wet Age-related Macular Degeneration in Italy
Brief Title: Aflibercept (Eylea) in roUtine Clinical Practice in patientS With Wet Age-related Macular Degeneration in Italy
Acronym: PERSEUS-IT
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Other Study IDs: 17634; EY1415IT (Other: Company Internal)
Record Dates: First submitted 2014-11-10; First posted 2014-11-13 (Estimated); Last update posted 2023-11-07 (Actual); Status verified 2023-11

CONDITIONS: Wet Macular Degeneration
Keywords: wet AMD
MeSH Terms: conditions — Wet Macular Degeneration | interventions — aflibercept

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Cohort 1: According to the recommendations of the Summary of Product Characteristics (SmPC) in Italy
  Interventions: Drug: Aflibercept (Eylea, VEGF Trap-Eye, BAY86-5321)

INTERVENTIONS:
Drug: Aflibercept (Eylea, VEGF Trap-Eye, BAY86-5321) — Administration by intravitreal injection

SUMMARY:
The main objectives of this non-interventional cohort field study are to evaluate effectiveness of Eylea and to describe follow-up as well as treatment patterns in patients with wAMD (wet age-related macular degeneration) in routine clinical practice in Italy for a study population of "naïve" patients

ELIGIBILITY:
Inclusion Criteria:

* "Naïve" patients with wet AMD(age-related macular degeneration) treated with Eylea (in accordance with the local Summary of Product Characteristics, SPC).

Exclusion Criteria:

* Exclusion criteria as listed in the local SPC. Scar, fibrosis, or atrophy involving the center of the fovea in the study eye.
* Any concomitant therapy with another agent to treat wet AMD in the study eye.
* Any prior or concomitant therapy with another drug for wAMD.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: wet AMD (wet age-related macular degeneration) patients
Sampling Method: Non-Probability Sample
Enrollment: 912 (Actual)
Dates: Start 2015-01-09 (Actual); Primary Completion 2019-03-28 (Actual); Study Completion 2019-07-08 (Actual)

PRIMARY OUTCOMES:
Mean change of visual acuity from baseline to 12 months. | Baseline to 12 months
Mean change of visual acuity from baseline to 24 months. | Baseline to 24 months

SECONDARY OUTCOMES:
Number of clinical visits (visits for injections) | At 12 and 24 months
Number of monitoring visits (visits only for diagnostic purposes, but without injections) | At 12 and 24 months
Number of combined visits (visits for monitoring and injection) | At 12 and 24 months
Number of post-injection monitoring visits (visits only for safety checks after injection) | At 12 and 24 months
Number of visits outside the study center after 12 and 24 months | At 12 and 24 months
Number of optical coherence tomography (OCT) assessments per patient | At 12 and 24 months
Number of visual acuity tests | At 12 and 24 months
Number of fundoscopy examinations | At 12 and 24 months
Mean time between the injections and visits | At 12 and 24 months
Mean time between the first symptoms and diagnosis | Up to 24 months
Mean time from indication of the Eylea treatment by the treating physician to treatment | Up to 24 months
  Time will be defined as difference in days between clinical indication for the treatment and the first injection
Proportion of patients with no fluid | At 4,12 and 24 months
Mean change in retinal thickness from baseline | Baseline and at 4,12 and 24 months
  As measured by OCT (SD-SLO) Optical Coherence Tomography ( Spectral Domain / Scanning Laser Ophthalmoscope)

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- Multiple Locations, Italy

REFERENCES:
- [Result] Nicolo M, Ciucci F, Nardi M, Parolini B, Russo A, Scupola A, Torregrossa S, Vadala M; PERSEUS-IT study investigators. PERSEUS-IT 24-month analysis: a prospective observational study to assess the effectiveness of intravitreal aflibercept in routine clinical practice in Italy in patients with neovascular age-related macular degeneration. Graefes Arch Clin Exp Ophthalmol. 2022 Oct;260(10):3185-3195. doi: 10.1007/s00417-022-05679-6. Epub 2022 May 5. PMID 35511286
- See also: Click here to find results for studies related to Bayer products — http://clinicaltrials.bayer.com/